CLINICAL TRIAL: NCT03494517
Title: Detection of Epileptiform Activity in Severe Preeclampsia: A Prospective Observational Pilot Study
Brief Title: Detection of Epileptiform Activity in Severe Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pascal Vuilleumier (Other)
Responsible Party: Sponsor-Investigator, Pascal Vuilleumier, Dr. Med., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: DEpiPre2018
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sFlt-1:PIGF ratio, LH, FSH, TSH, fT4, Oestradiol (E2), Progesterone. Magnesium levels after 4 hours of infusion (steady state), 48 and 72h.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preeclampsia: Women aged 18-45 years
  1. Confirmed pregnancy > 30 weeks of gestation
  2. Singleton or multiple pregnancies
  3. Admission in maternity of the Women's hospital with clinically suspected signs of severe preeclampsia:
     * Systolic blood pressure >140 mmHg or diastolic pressure > 90 mmHg and
     * Proteinuria > 0.3 grams in a 24-hour urine or protein:creatinine ratio >0.3 or
     * Signs of end-organ dysfunction (platelet count < 100'000G/l, serum creatinine >110 mg/l, or doubling of the serum creatinine, elevated serum transaminases to twice normal concentration)
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Baseline EEG measurement will be performed for 5 minutes before intravenous magnesium administration will start as defined by the administration scheme of the Women's Hospital of the Bern University Hospital. After completion of the bolus infusion and at the beginning of the maintenance infusion of magnesium the second EEG measure will be performed for another 5 minutes. After 4 hours of intravenous magnesium treatment the plasmatic magnesium concentration is expected to be at a steady-state. A third 5-minute measure will be performed at this time point.

SUMMARY:
The primary aim of this pilot study is to prospectively quantify epileptiform activity in a cohort of preeclamptic patients before and after intravenous magnesium administration.

Secondary aims will be the exploration of a potential association between epileptiform activity and the sFlt-1:PIGF ratio, as well as a correlation to clinical signs of preeclampsia.

A positive finding may aid obstetricians to detect an increased convulsive risk by performing a simplified EEG early in the diagnostic path of preeclampsia. If confirmed in a larger trial positive correlations of an increased sFlt-1:PIGF ratio with epileptiform activity might be a risk marker for early severe preeclampsia, guiding obstetricians into clinical decision-making in regard to an increased maternal risk of eclampsia.

DETAILED DESCRIPTION:
Preeclampsia constitutes a heterogeneous multisystemic disorder defined by the new onset of hypertension and proteinuria after 20 weeks of gestation.1 The incidence of preeclampsia in Switzerland is estimated at 2.31 % of pregnancies (95% CI 1.62-3.28%), about 1'911 cases/year can be expected to occur on the national level. Preeclampsia and eclampsia are considered a continuum in the hypertensive disorders of pregnancy. When convulsions or coma occur in addition to hypertension the condition is referred to as eclampsia. Up to 2-3% of severely preeclamptic women will have eclampsia,4 with a consecutive mortality rated between 0-14%.5 The diagnosis of preeclampsia is challenging, because of clinical heterogenity, especially at early stages. Until recently no routine laboratory test or biological marker other than presenting clinical symptoms such as severe headache or arterial hypertension, decreased plasmatic thrombocyte count and proteinuria were available for diagnostic purposes.

The only curative treatment of severe preeclampsia and eclampsia consists of delivery of fetus and placenta. Since the 2002 Magpie trial, the mainstay of eclampsia prevention in severely preeclamptic patients relies on the prophylactic use of intravenous magnesium, either when prompt delivery can be performed, or if it has to be delayed for fetal reasons. Obviously, eclampsia prevention is critical, considering that eclampsia onset can occur pre, intra, or postpartum. Hereby the prophylactic magnesium treatment is mostly maintained throughout a period of several days before and after delivery of the fetus and placenta, as up today there is no reliable clinical or diagnostic approach to predict the risk of eclamptic seizures.

The actual gold standard in high-risk maternities is to assess clinical symptoms as described above and perform newer laboratory essays, in order to estimate the parturient's risk for preeclamptic complications. Insofar changes in serum levels of fms-like tyrosine kinase-1 (sFlt-1) and placental growth factor (PGIF) were lately revealed and have been currently approved as diagnostic aid in preeclampsia. Circulating maternal serum levels of sFlt-1 are increased, and PGIF are decreased in preeclampsia. As an antagonist of PGIF and vascular endothelial growth factor, sFlt-1 causes vasoconstriction and endothelial damage. Noteworthy a sFlt-1:PIGF ratio lower than 38 can be used as to predict a short-term absence of preeclampsia in women with suspect clinical symptoms.

Interestingly novel knowledge points to a strong link in between plasmatic steroid hormones and epilepsy, with strong animal data pointing towards a higher epileptogenic potential in high estrogenic states; whereas androgens, namely progesterone seem to induce a protective state through agonism on extrajunctional GABAA receptors.

EEG slopes are good markers for epileptiform activity. EEG changes have been reported in eclampsia and in severe preeclampsia, with differences also reported between severe preeclampsia and eclampsia.Recently, slow waves most frequently localized in the occipital lobe, as well as spike discharges in EEG, were reported as warning signs of deterioration of brain function in preeclampsia or eclampsia. Neither have electroencephalic correlates of sFlt-1, PGIF or hormonal states been investigated in preeclampsia. EEG is not in routine use for convulsive risk assessment in maternity wards, when preeclampsia screening is performed. One of the reasons might be that performing EEGs is time consuming and involves significant human resources for urgent EEG analysis. These resources might be lacking even in tertiary hospitals. Novel reliable, noninvasive and technically easy to perform simplified EEG methods have become available, these are especially in use during anesthesia for detection of clinically silent epileptic potentials.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed pregnancy > 30 weeks of gestation
2. Singleton or multiple pregnancies
3. Admission in maternity of the Women's hospital with clinically suspected signs of severe preeclampsia:

   * Systolic blood pressure >140 mmHg or diastolic pressure > 90 mmHg and
   * Proteinuria > 0.3 grams in a 24-hour urine or protein:creatinine ratio >0.3 or
   * Signs of end-organ dysfunction (platelet count < 100'000G/l, serum creatinine >110 mg/l, or doubling of the serum creatinine, elevated serum transaminases to twice normal concentration)

Exclusion Criteria:

1. Lack of patient's informed consent
2. Active labor
3. Eclampsia
4. Hypertensive crisis as defined by Systolic blood pressure > 210 mmHg or diastolic pressure > 120 mmHg
5. Known epilepsy
6. Posterior reversible encephalopathy syndrome
7. Antiepileptic medication (except magnesium sulfate)
8. Reported or admitted medication or substance abuse (street drugs, opiates, benzodiazepines, alcohol)
9. Known neurologic condition with previously pathologic diagnostic imaging or EEG
10. Severe fetal malformations (abdominal: gastroschisis & omphalocele, tracheoesophageal fistula, cerebral: brain malformations included in the category of cephalic disorders, pulmonary: lung hypoplasia, cardiac: congenital heart disease)
11. Preceding rupture of membranes
12. Non-German and non-French speaking parturient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Preeclampsia in pregnant women
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Epileptiform activity | 0-4h after Magnesium Sulfate administration
  The primary aim of this pilot study is to prospectively quantify epileptiform activity in a cohort of preeclamptic patients before and after intravenous magnesium administration. Analysis of the EEG will include baseline spectral analysis (e.g. density spectral array), but the main focus will be the detection of epileptiform signals by absolute slope and ordinal pattern analysis.

SECONDARY OUTCOMES:
Biological correlates to epileptiform activity | 72h after inclusion
  Secondary aims will be the exploration of a potential association between epileptiform activity and the sFlt-1:PIGF ratio, as well as a correlation to clinical signs of preeclampsia.
  Screening for epileptic potentials will be performed by absolute slope analysis on the EEG. EEG data will be used as categorical variables (yes/no potentials), thereafter by logistic regression and propensity matching concerning the association between the baseline amount of EEG abnormality and plasma values of sFlt-1:PGIF-ratio.
Demographics of mother and infant | 72h after inclusion
  Mother: Age, gender, weight and body-mass-index, diabetes or gestational diabetes mellitus, antihypertensive medication, anticoagulant and antiplatelet treatment, mode of delivery, drugs administered at admission, after 4, 6, 12, 24, 48 and 72h, clinical outcome.
  Infant: Weeks of gestation, weight, 5 min. APGAR, cord pH at birth, transfer to neonatal intensive care unit, meconium aspiration syndrome, respiratory distress syndrome and neonatal sepsis.
  Maternal laboratory measures: At admission: sFlt-1:PIGF ratio, LH, FSH, TSH, fT4, Oestradiol (E2), Progesterone. Magnesium levels after 4 hours of infusion (steady state), 48 and 72h.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal H Vuilleumier, MD, Principal Investigator — Bern University Hospital
Locations (1):
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD will remain within a secured server (Labkey) and will only be shared to the study officials for analysis purposes.